CLINICAL TRIAL: NCT02763124
Title: Pseudophakic Astigmatic Reduction With Verion-LenSx Arcuate Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Alcon, a Novartis Company (Industry)
Responsible Party: Principal Investigator, Clayton Blehm, MD, PI, Gainesville Eye Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-16-001
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Astigmatism
Keywords: Pseudophakic
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Verion-LenSx (Experimental): The Verion-LenSx femtosecond laser system will be used to perform one or two corneal arcuate incisions.
  Interventions: Procedure: Verion-LenSx

INTERVENTIONS:
Procedure: Verion-LenSx — The Verion-LenSx femtosecond laser system will be used to create one or two partial-depth corneal arcuate incisions

SUMMARY:
To assess the effectiveness of the Verion-LenSx guided arcuate incision technique to reduce astigmatism in a pseudophakic population.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of corneal arcuate incisions when they are performed with a femtosecond laser system on subjects who have had previous cataract surgery. The procedure to be used would not be different from that employed during cataract surgery, except that the only corneal incisions made would be the partial-depth arcuate incisions at the laser.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or older
* Willing and able to provide informed consent for participation in the study.

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Verion-LenSx
Started | 18; 28 Eyes
Completed | 18; 28 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Verion-LenSx
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.1)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 19
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Refractive cylinder (diopters) [Mean (Standard Deviation); unit: diopters] | 1.35 (0.30)
Average keratometry (diopters) [Mean (Standard Deviation); unit: diopters] | 44.27 (1.41)
Corneal astigmatism (diopters) [Mean (Standard Deviation); unit: diopters] | 1.42 (.54)

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Monocular Distance Visual Acuity
Description: Uncorrected monocular distance visual acuity, measured on a logMAR scale, (logarithm of the Minimum Angle of Resolution) which is a measure of visual acuity in which the smaller values indicate better visual acuity.
Time Frame: 60 days (+/- 10 days) after laser treatment
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Verion-LenSx
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 28
logMAR | 0.14 (0.11)

2. Secondary Outcome: Change in Corneal Astigmatism
Description: Vector change in the astigmatism measured on the cornea, in diopters
Time Frame: 60 days (+/- 10 days) after laser treatment
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Verion-LenSx
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 28
diopters | 1.2 (0.74)

3. Secondary Outcome: Change in Refractive Cylinder
Description: The vector change in refractive cylinder in diopters
Time Frame: 60 days (+/- 10 days) after laser treatment
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Verion-LenSx
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 28
diopters | 1.21 (0.42)

4. Secondary Outcome: Spectacle Independence at Distance
Description: Percentage of subjects that do not rely on spectacles for distance vision
Time Frame: 60 days (+/- 10 days) after laser treatment
Population: There were 28 eyes of 18 subjects treated in the study. Spectacle independence is evaluated by subject, not eye.
Measure: Count of Participants; unit: Participants
Arm/Group | Verion-LenSx
Number analyzed (Participants) | 18
Participants | 12

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | Verion-LenSx
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verion-LenSx (N=18)
Corneal ulcer (Eye disorders) | 1 (1) — Corneal ulcer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes